CLINICAL TRIAL: NCT00473174
Title: A Prospective, Randomized, Open Label, Blinded-endpoint Study to Compare Awakening Versus Bedtime Administration of 5-10 mg Ramipril in Terms of Systolic Blood Pressure Lowering Determined by ABPM in Subjects With Mild-to-moderate Essential
Brief Title: Comparison of Awakening Versus Bedtime Dosing of Ramipril in Subjects With Essential Hypertension
Acronym: HYCCRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Ramon C. Hermida, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYCCRA-2006/01; Eudract-2006-006107-37
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Hypertension
Keywords: Ramipril; Ambulatory blood pressure monitoring; Chronotherapy; Circadian; Non-dipper
MeSH Terms: conditions — Hypertension | interventions — Ramipril; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ramipril on awakening
  Interventions: Drug: Ramipril; Device: ambulatory blood pressure monitoring
- 2 (Active Comparator): Ramipril at bedtime
  Interventions: Drug: Ramipril; Device: ambulatory blood pressure monitoring

INTERVENTIONS:
Drug: Ramipril — Dosing on awakening versus bedtime
Device: ambulatory blood pressure monitoring — Blood pressure measured at 20-min intervals from 07:00 to 23:00 hours and at 30-min intervals at night for 48 consecutive hours

SUMMARY:
This prospective chronotherapy trial will investigate the potential differing efficacy of ramipril in doses from 5 to 10 mg/day when administered, as a monotherapy either upon awakening from nighttime sleep or at bedtime, to diurnally active patients with grade 1 or 2 essential hypertension, who will be evaluated by 48-hour ABPM before and after pharmacologic intervention. The benefits from this trial may be extremely important, taking into account

1. the high prevalence of non-dipping among patients with essential hypertension
2. the need for a proper 24-hour BP control with particular emphasis on the regulation of nighttime resting BP mean
3. the lacking information on the administration-time dependent effects on BP of ramipril, a widely used ACEI in doses of 5-10 mg/day.

DETAILED DESCRIPTION:
Several attributes of the cardiovascular system, including blood pressure (BP) and heart rate (HR), are characterized by predictable changes during the 24 hours for the most part in synchrony with the rest-activity cycle. During the past two decades specific features of the 24-hour BP pattern have been assessed as potential sources of injury to target tissues and as triggers of cardiac and cerebrovascular events in hypertensive patients. A growing number of studies indicate the reduction of the normal 10 to 20% sleep-time BP decline (non-dipper pattern) is associated with elevated risk of end-organ injury, particularly to the heart (left ventricular hypertrophy and myocardial infarct), brain (stoke) and kidney (albuminuria and progression to end-stage renal failure). Accordingly, there is growing interest in how to tailor the treatment of hypertensive patients according to their circadian BP pattern.

Clinical studies demonstrated a different effect of the ACEIs benazepril, enalapril, perindopril, quinapril, spirapril, and trandolapril when dosed in the morning versus the evening. A small trial on 33 patients with essential hypertension showed that a low dose of 2.5 mg/day ramipril more effectively reduced daytime BP when it was administered in the morning and more effectively reduced nighttime BP when it was administered in the evening. In the HOPE (Heart Outcomes Prevention Evaluation) study patients in the active treatment group received ramipril at bedtime. Results from a small substudy, in which hypertensive patients were evaluated with 24-hour ambulatory BP monitoring (ABPM), showed a marked BP reduction particularly during nighttime sleep, thereby reducing the prevalence of non-dippers. The authors concluded that the effects on cardiovascular morbidity and mortality seen with ramipril in the HOPE study may relate to its improved effect (i.e., increase in the diurnal/nocturnal BP ratio) on the non-dipping BP patterns.

In keeping with the documented administration-time dependent effects on BP regulation of other ACEI, this prospective chronotherapy trial will investigate the potential differing efficacy of ramipril in doses from 5 to 10 mg/day when administered, as a monotherapy either upon awakening from nighttime sleep or at bedtime, to diurnally active patients with grade 1 or 2 essential hypertension, who will be evaluated by 48-hour ABPM before and after pharmacologic intervention. The benefits from this trial may be extremely important, taking into account 1) the high prevalence of non-dipping among patients with essential hypertension, 2) the need for a proper 24-hour BP control with particular emphasis on the regulation of nighttime resting BP mean, and 3) the lacking information on the administration-time dependent effects on BP of ramipril, a widely used ACEI in doses of 5-10 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension

Exclusion Criteria:

* Severe hypertension.
* Secondary hypertension.
* Grade III/IV hypertensive retinopathy.
* Type 1 diabetes.
* Cerebrovascular or cardiovascular event during the last 12 months prior to inclusion.
* Pregnant or lactating females.
* History of malignancy within the past five years.
* Shift workers.
* Obstructive sleep apnea.
* Use of disallowed concomitant medication.
* Intolerant to ABPM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of bedtime administration of ramipril in subjects with essential hypertension by testing the hypothesis of superior nocturnal SBP lowering in ABPM measurements compared with ramipril administered on awakening | Three months

SECONDARY OUTCOMES:
To demonstrate that ramipril at bedtime is more effective than ramipril upon awakening in terms of nocturnal DBP lowering in ABPM | Three months
To demonstrate that ramipril at bedtime is not inferior to ramipril upon awakening in terms of 24-hour SBP/DBP lowering in ABPM | Three months
To demonstrate that ramipril at bedtime is more effective than ramipril upon awakening in terms of increasing the diurnal/nocturnal SBP and DBP ratio determined by ABPM | Three months
To demonstrate that ramipril at bedtime offers a similar safety profile than ramipril upon awakening | Three months
To demonstrate that compliance with ramipril at bedtime is similar to compliance of ramipril upon awakening | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, PhD, Principal Investigator — University of Vigo
Locations (1):
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, Spain

REFERENCES:
- [Result] Hermida RC, Ayala DE. Chronotherapy with the angiotensin-converting enzyme inhibitor ramipril in essential hypertension: improved blood pressure control with bedtime dosing. Hypertension. 2009 Jul;54(1):40-6. doi: 10.1161/HYPERTENSIONAHA.109.130203. Epub 2009 May 11. PMID 19433778